CLINICAL TRIAL: NCT04722757
Title: Functional Outcomes of Transanal Ileal Pouch-Anal Anastomosis Compared to Laparoscopic or Open Ileal Pouch-Anal Anastomosis: a Multi-Center, Randomized, Parallel-Group, Non-Inferiority Trial
Brief Title: Comparison of Functional Outcomes Between Transanal and Laparoscopic vs Open Ileal Pouch-Anal Anastomosis
Acronym: FUNCTIon
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Cedars-Sinai Medical Center (Other); St Mary's Hospital, London (Other); Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Anthony DeBuck, Assistant Professor, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-0260-A
Record Dates: First submitted 2021-01-20; First posted 2021-01-25 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Ulcerative Colitis; Inflammatory Bowel Diseases; Ileal Pouch
Keywords: transanal surgery, pouch function
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: The FUNCTIon trial is designed as a multicenter, open-label, 2-arm parallel-group, non-inferiority randomized multicenter international trial. Randomization will be stratified by center, with permuted blocks and balanced allocation (1:1). Neither participants nor treating physicians will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transanal IPAA (Experimental): In the experimental arm, patients will undergo transanal dissection of the distal part of the rectum. After proctectomy, an ileal pouch-anal anastomosis (IPAA) will be created. A Gelpoint Path will be used to create access through the anus. Postoperative care will occur following the hospital specific protocols.
  Interventions: Procedure: ta-IPAA
- transabdominal IPAA (Active Comparator): In the control group, proctectomy will occur through abdominal dissection (laparoscopy, single port laparoscopy, robotic or open). Postoperative care will occur following the hospital specific protocols.
  Interventions: Procedure: tabd-IPAA

INTERVENTIONS:
Procedure: ta-IPAA — A trans-anal port (gelpoint path, Applied Medical®) will be used for transanal acces and pneumopelvis will be created. The initial purse string is to be placed approximately 3cm above the dentate line, followed by a rectotomy. The perirectal dissection is then continued and should be pursued for at least 5cm. More proximal dissection can be done by transabdominal access. After completion of the proctectomy, a double purse string anastomosis is performed after creation of the J-pouch. A defunctioning loop ileostomy can be placed according to surgeon's preference.
  Arms: transanal IPAA
Procedure: tabd-IPAA — Patients in the control group will undergo a rectal dissection by laparotomy, Pfannenstiel incision, (hand-assisted) laparoscopy, single port laparoscopy or robotic surgery, but performed from the abdominal side (tabd-IPAA). Dissection will be performed down to the pelvic floor and include the distal rectum. It is anticipated that most dissection will occur using the TME plane, however, close rectal dissection is also acceptable. Transection of the distal rectum approximately 2 cm above the dentate line will be performed using a linear stapler of the surgeon's choice. After placing the anvil in the J-pouch, a circular stapler will be introduced through the sphincter and a circular anastomosis will be performed. A defunctioning loop ileostomy can be placed according at the surgeon's discretion.
  Arms: transabdominal IPAA

SUMMARY:
Background: Ulcerative colitis (UC) and inflammatory bowel unclassified (IBDu) are inflammatory bowel diseases (IBD) involving the colon and rectum. It is a chronic disease occurring in young people with a high burden on social and professional life. Although treated medically by immunomodulatory drugs, about 15 - 20% of UC patients will need an ileal pouch-anal anastomosis (IPAA). In primary cases, this procedure is usually performed laparoscopically (further called transabdominal IPAA or tabd-IPAA). More recently even less invasive surgical techniques have emerged, using a trans-anal access, facilitating dissection of the distal rectum. Although transanal access is associated with a good postoperative outcome profile, there is very limited data on functional outcome in patients with a trans-anal ileal pouch-anal anastomosis surgery (ta-IPAA).

Objective: The objective of this study is to determine if functional outcome following ta-IPAA is the same as or better than postoperative function after tabd-IPAA with UC and IBDu.

Study design: The FUNCTIon trial is a non-inferiority randomized, controlled trial that will involve 3 hospitals across North-America and Europe.

Patient population: All patients with UC and IBDu eligible for pelvic pouch procedure will be randomized to either ta-IPAA or tabd-IPAA. Prior to the start of the study REB will be obtained at all centres and informed consent will be obtained from all patients. The inclusion criteria for the study are: patients between 18 and 60 years old with UC or IBD unclassified (IBDu) eligible for surgery. They will need to speak either English or the primary language of the center they are treated at. The exclusion criteria for the study are: contraindication for laparoscopy, familial adenomatous polyposis (FAP), colorectal cancer, presence of primary sclerosing cholangitis (PSC), a hand-sewn ileo-anal anastomosis, immunomodulating therapy including steroids, pregnancy and lactating, urgent indication.

Intervention: ta-IPAA or tabd-IPAA. Outcomes: Primary outcome is the functional outcome at one year after pelvic pouch surgery. This will be measured using the validated Colorectal Functional Outcome (COREFO) questionnaire. Secondary outcomes are functional outcome at 3 and 6 months, male and female sexual function, perioperative measures and clinical measures.

Sample Size: A sample of 48 (24 per group) is required to detect a between-group non-inferiority margin of 7.05 in COREFO score with a 1-sided α of 0.05 and a power of 80%, allowing for 20% attrition. A participation rate of 50% is anticipated.

Analysis: All continuous variable outcomes will be compared using analysis of covariance. Categorical variable outcomes will be analyzed using repeated measures logistic regression. Proportional outcomes will be analyzed with the chi-square or Fisher's exact test and continuous variables will be analyzed with student's t-test.

Follow-up: Each participant will be followed up at 6 weeks, 3 months, 6 months and 12 months after the intervention to assess functional scores and clinical events. Perioperative events (including postoperative complications) will be assessed during the intervention hospitalization period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with UC or IBD-U refractory to medical therapy or with dysplasia
2. Patients undergoing a 1-, 2-stage, 3-stage approach
3. Between 18 years old and 60 years old.
4. Speak English and/or primary language of recruiting center.
5. Provide informed consent

Exclusion Criteria:

1. Patients with familial adenomatous polyposis (FAP);
2. Patients with contraindications for laparoscopic surgery including previous laparotomy, toxic megacolon and chronic obstructive pulmonary disease (COPD) Gold III or higher;
3. Patients still taking steroids at the time of proctectomy and IPAA construction. A wash-out period of 8 weeks will be considered for all treatments before performing the pouch construction.
4. Patients with confirmed or suspected colorectal cancer;
5. Patients with primary sclerosing cholangitis (PSC)
6. Patients needing a hand-sewn anastomosis;
7. Redo-pouch surgery
8. Pregnancy and lactation (tested by a urinary pregnancy test)
9. Patients undergoing an urgent or emergent proctocolectomy. Those patients are still eligible if they undergo a subtotal colectomy first and a completion proctectomy in a second stage.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Pouch function | 12 months after pouch construction or stoma closure
  The primary outcome measure is the difference in functional outcome between the ta-IPAA and tabd-IPAA, measured by the Colorectal Functional Outcome (COREFO) questionnaire at 12 months after pouch surgery. Since this is a non-inferiority study, the hypothesis is that functional outcome 12 months after ta-IPAA is not worse than after tabd-IPAA. COREFO is a validated functional score used to assess colorectal function, divided in 5 domains (Incontinence, social impact, frequency, stool related aspects and need for medication) with a total of 27 questions and a result expressed between 0 and 100, increasing with a worse function.

SECONDARY OUTCOMES:
Pouch function | 3 and 6 months after pouch construction or stoma closure
  Colorectal Functional Outcome (COREFO). The score ranges between 0 and 100, increasing with a worse function
Anastomotic Leak Rate | 6 weeks after pouch construction
  Diagnostic assessment will occur by either a contrast enema or CT with both intravenous contrast and anal contrast enema in patients in which leaks are clinically suspected. In defunctioned pouches, a contrast enema will be performed before stoma closure. This will be organized at 6 weeks.
Postoperative Morbidity | 30 days after pouch construction
  Thirty-day morbidity of the index surgery will be reported and expressed using the Dindo-Clavien classification. The main advantage of this scoring system is that it takes all complications into account instead of considering only the most severe complication.
Readmission | 30-day after pouch construction
  Readmission to hospital
Patient's Quality of Life | 3,6 and 12 months after pouch construction
  Patient-Reported Outcomes Measurement Information System Global Health (PROMIS GLOBAL-10)
Sexual function | 3,6 and 12 months after pouch construction
  Patient-Reported Outcomes Measurement Information System Sexual Function and Satisfaction (PROMIS-SexFS)
Urinary Function | 3,6 and 12 months after pouch construction
  International Prostate Symptom Score (IPSS). The score ranges between 1 and 35, increasing with a worse symptom (Mild: 1-7, Moderate: 8-19, Severe: 20-35)
Fecal Incontinence | 3,6 and 12 months after pouch construction
  Wexner incontinence score. The score ranges between 0 and 20, where 0 is perfect continence and 20 is complete incontinence.

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided